CLINICAL TRIAL: NCT02595983
Title: An Open-label Study to Evaluate the Efficacy and Safety of Revusiran in Patients With Transthyretin-mediated Familial Amyloidotic Polyneuropathy With Disease Progression Post-Orthotopic Liver Transplant
Brief Title: The Study of an Investigational Drug, Revusiran (ALN-TTRSC), for the Treatment of Transthyretin (TTR)-Mediated Amyloidosis in Patients Whose Disease Has Continued to Worsen Following Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTRSC-005
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Results first posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Transthyretin (TTR)-Mediated Amyloidosis; Familial Amyloidotic Polyneuropathy (FAP); ATTR Amyloidosis; Familial Amyloid Neuropathies
Keywords: FAP; Familial Amyloidotic Polyneuropathy; ATTR Amyloidosis; Orthotopic Liver Transplant; RNAi therapeutic
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — revusiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): All patients who received at least 1 dose of revusiran (ALN-TTRSC)
  Interventions: Drug: Revusiran

INTERVENTIONS:
Drug: Revusiran — 500mg Revusiran by subcutaneous (sc) injection
  Other Names: ALN-TTRSC

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of revusiran (ALN-TTRSC) in adults with transthyretin-mediated amyloidosis (ATTR), whose disease has continued to worsen after liver transplantation. Dosing has been discontinued; patients are being followed-up for safety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FAP (familial amyloidotic polyneuropathy) with documented TTR mutation
* Received an orthotopic liver transplant ≥12 months before the date of informed consent
* An increase in polyneuropathy disability (PND) score post-transplant
* Polyneuropathy Disability score of ≤3b

Exclusion Criteria:

* New York Heart Association (NYHA) classification of >2
* Other known causes of sensorimotor or autonomic neuropathy (eg, autoimmune disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Vest, MD, Study Director — Alnylam Pharmaceuticals
Locations (6):
- Clinical Trial SIte, Paris, France
- Clinical Trial SIte, Münster, Germany
- Clinical Trial SIte, Porto, Portugal
- Clinical Trial SIte, Majorca, Spain
- Clinical Trial Site, Umeå, Sweden
- Clinical Trial SIte, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants with hereditary Transthyretin-mediated Amyloidosis (ATTR) with polyneuropathy who had neuropathy progression following post-orthotopic liver transplant (OLT) were enrolled and treated in this study.
Groups:
- All Patients: All patients who received at least 1 dose of revusiran
Period: Overall Study
Arm/Group | All Patients
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Familial Amyloidotic Polyneuropathy (FAP) Stage [Count of Participants; unit: Participants]
  FAP Stage I: Unimpaired ambulation | 3
  FAP Stage II: Assistance with ambulation required | 9
  FAP Stage III: Wheelchair-bound or bedridden | 0
Serum Transthyretin (TTR) [Mean (Standard Deviation); unit: micrograms/milliliter (μg/mL)] | 192.3 (43.28)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Serum TTR at Month 6
Description: A negative percentage change from baseline at Month 6 indicates a reduction in serum TTR level.
Time Frame: Month 6
Population: Safety analysis set: All participants who received at least a single dose of study drug and for whom data were collected at Month 6.
Measure: Mean (Standard Deviation); unit: percentage change from baseline in TTR
Groups:
- All Patients: All patients who received at least 1 dose of study drug
Arm/Group | All Patients
Number analyzed (Participants) | 7
percentage change from baseline in TTR | -72.0 (18.39)

2. Secondary Outcome: Percentage Change From Baseline in Serum TTR Over 18 Months
Description: A negative percentage change from baseline indicates a reduction in serum TTR level.
Time Frame: Weeks 3, 7, 12, 18, 24, 26 (Month 6), 39 (Month 9), 52 (Month 12), 57, 78 (Month 18)
Population: Safety analysis set: All participants who received at least a single dose of study drug and for whom data were collected at each time point. Data collection was limited due to the discontinuation of the drug treatment early in the study as per protocol amendment.
Measure: Mean (Standard Deviation); unit: percentage change from baseline in TTR
Arm/Group | All Patients
Number analyzed (Participants) | 12
percentage change from baseline in TTR
  Week 3 | -75.1 (18.79)
  Week 7 | -79.0 (15.46)
  Week 12 | -73.0 (18.61)
  Week 18: number analyzed (Participants) | 10
  Week 18 | -73.5 (14.30)
  Week 24: number analyzed (Participants) | 8
  Week 24 | -73.4 (14.32)
  Week 26 (Month 6): number analyzed (Participants) | 7
  Week 26 (Month 6) | -72.0 (18.39)
  Week 39 (Month 9): number analyzed (Participants) | 0
  Week 52 (Month 12): number analyzed (Participants) | 0
  Week 57: number analyzed (Participants) | 0
  Week 78 (Month 18): number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Modified Neurological Impairment Score (mNIS +7) Composite Score Over 18 Months
Description: The mNIS+7 is a composite score that measures neurologic impairment which includes the following components: physical exam of lower limbs, upper limbs and cranial nerves to assess motor strength/weakness, electrophysiologic measurement of small and large nerve fiber function, sensory testing and postural blood pressure. The minimum and maximum values are 0 and 304, respectively. A higher score indicates a worse outcome. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Months 6, 12, 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 12
score on a scale
  Baseline | 90.4 (43.76)
  Change from baseline at Month 6: number analyzed (Participants) | 7
  Change from baseline at Month 6 | 6.9 (10.42)
  Change from baseline at Month 12: number analyzed (Participants) | 0
  Change from baseline at Month 18: number analyzed (Participants) | 0

4. Secondary Outcome: Norfolk Quality of Life-Diabetic Neuropathy (QoL-DN) Questionnaire Score
Description: The Norfolk QoL-DN questionnaire is a standardized 35-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy - small fiber, large fiber, and autonomic nerve function. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
Time Frame: Baseline, Months 6, 12, 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 12
score on a scale
  Baseline | 61.3 (24.86)
  Month 6: number analyzed (Participants) | 7
  Month 6 | 77.1 (31.06)
  Month 12: number analyzed (Participants) | 0
  Month 18: number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants in Each Polyneuropathy Disability (PND) Stage Based on Worst Post-Baseline Score
Description: PND Scores: Stage 0: No symptoms, Stage 1: Sensory disturbances but preserved walking capabilities, Stage 2: Impaired walking capacity, but ability to walk without a stick or crutches, Stage 3A/B: Walking with help of 1 or 2 sticks or crutches, Stage 4: confined to wheel chair. For each stage (0-4) at baseline, the number of participants is presented at their worst post-baseline score for each stage (0-4) post-baseline. Worst post-baseline is defined the highest PND classification for a participant recorded after the first dose of study drug.
Time Frame: Baseline, Months 6, 12, 18
Population: Safety analysis set: All participants who received at least a single dose of study drug and for whom data were collected post-baseline. Data collection was limited due to the discontinuation of the drug treatment early in the study as per protocol amendment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 11
Participants
  Baseline Stage 0, Post-baseline Stage 0 | 0
  Baseline Stage 0, Post-baseline Stage 1 | 0
  Baseline Stage 0, Post-baseline Stage 2 | 0
  Baseline Stage 0, Post-baseline Stage 3A/B | 0
  Baseline Stage 0, Post-baseline Stage 4 | 0
  Baseline Stage 1, Post-baseline Stage 0 | 0
  Baseline Stage 1, Post-baseline Stage 1 | 1
  Baseline Stage 1, Post-baseline Stage 2 | 0
  Baseline Stage 1, Post-baseline Stage 3A/B | 0
  Baseline Stage 1, Post-baseline Stage 4 | 0
  Baseline Stage 2, Post-baseline Stage 0 | 0
  Baseline Stage 2, Post-baseline Stage 1 | 1
  Baseline Stage 2, Post-baseline Stage 2 | 0
  Baseline Stage 2, Post-baseline Stage 3A/B | 0
  Baseline Stage 2, Post-baseline Stage 4 | 0
  Baseline Stage 3A/B, Post-baseline Stage 0 | 0
  Baseline Stage 3A/B, Post-baseline Stage 1 | 0
  Baseline Stage 3A/B, Post-baseline Stage 2 | 1
  Baseline Stage 3A/B, Post-baseline Stage 3A/B | 6
  Baseline Stage 3A/B, Post-baseline Stage 4 | 2
  Baseline Stage 4, Post-baseline Stage 0 | 0
  Baseline Stage 4, Post-baseline Stage 1 | 0
  Baseline Stage 4, Post-baseline Stage 2 | 0
  Baseline Stage 4, Post-baseline Stage 3A/B | 0
  Baseline Stage 4, Post-baseline Stage 4 | 0

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred after the start of study drug administration on Day 0 (Baseline) up to 90 days post modified early termination visit (End of Study)
Description: The same event may appear as both an AE and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study
Groups:
- Safety Population: All patients who received at least 1 dose of revusiran
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=12)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Death (General disorders) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Urinary tract infections (Infections and infestations) | 1 (2)
Blood immunoglobulin M increased (Investigations) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Adrenal adenma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Hypercapnic Coma (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=12)
Oedema peripheral (General disorders) | 4 (6)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (5)
Renal Failure (Renal and urinary disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (4)
Marcocytosis (Blood and lymphatic system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (4)
Urinary tract infection (Infections and infestations) | 2 (4)
Cardiac Failure (Cardiac disorders) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Injection Site Erythema (General disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Injection site haematomia (General disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalized Oedema (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Secretion discharge (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Prothrombin level decreased (Investigations) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1)
Blood pyruvic acid increased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eschar (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Blood pressure abnormal (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dosing of participants was discontinued early in this study and a protocol amendment allowed additional safety follow-up visits. This study completed based on the amendment, but only a limited amount of data was collected in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT02595983/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT02595983/SAP_001.pdf